CLINICAL TRIAL: NCT04333420
Title: A Pragmatic Adaptive Randomized, Controlled Phase II/III Multicenter Study of IFX-1 in Patients With Severe COVID-19 Pneumonia
Brief Title: Randomized, Controlled Study of IFX-1 in Patients With Severe COVID-19 Pneumonia
Acronym: PANAMO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IFX-1-P2.9; 2020-001335-28 (EudraCT Number)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Results first posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-03

CONDITIONS: Severe COVID-19 Pneumonia
Keywords: COVID-19 related severe pneumonia
MeSH Terms: interventions — vilobelimab; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two phases with 2 parallel arms each
Who Masked: Participant, Investigator
Masking Description: Phase II: Open label study (30 patients), Phase III: Double- blind (360 patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase II: IFX-1 + BSC (Experimental): Phase II study part: IFX-1: 800mg intravenously administered, BSC: Best supportive care
  Interventions: Drug: IFX-1 + BSC
- Phase II: BSC (Other): Phase II study part: BSC: Best supportive care
  Interventions: Drug: BSC
- Phase III: IFX-1 + SOC (Experimental): Phase III study part: IFX-1: 800mg intravenously administered, SOC: Standard of care
  Interventions: Drug: IFX-1 + SOC
- Phase III: Placebo + SOC (Placebo Comparator): Phase III study part: Placebo: placebo infusion intravenously administered, SOC: Standard of care
  Interventions: Drug: Placebo + SOC

INTERVENTIONS:
Drug: IFX-1 + BSC — Phase II study part: IFX-1 + BSC
  Other Names: Vilobelimab + Best Supportive Care
  Arms: Phase II: IFX-1 + BSC
Drug: BSC — Phase II study part: BSC
  Other Names: Best Supportive Care
  Arms: Phase II: BSC
Drug: IFX-1 + SOC — Phase III study part: IFX-1 + SOC
  Other Names: Vilobelimab + Standard of Care
  Arms: Phase III: IFX-1 + SOC
Drug: Placebo + SOC — Phase III study part: Placebo + SOC
  Other Names: Placebo + Standard of Care
  Arms: Phase III: Placebo + SOC

SUMMARY:
Phase II & Phase III:

This is a pragmatic, adaptive, randomized, multicenter phase II/III study evaluating IFX-1 for the treatment of COVID-19 related severe pneumonia. The study consists of two parts: Phase II, an open-label, randomized, 2-arm phase evaluating best supportive care (BSC) + IFX-1 (Arm A) and BSC alone (Arm B); and Phase III, a double-blind, placebo-controlled, randomized phase comparing standard of care (SOC) + IFX-1 (Arm A) versus SOC + placebo-to-match (Arm B)

DETAILED DESCRIPTION:
The phase II and Phase III portions enrolled patients subsequently.

1st patient was enrolled in the phase III portion on 1st October 2020.

ELIGIBILITY:
Phase II

Inclusion Criteria:

* At least 18 years of age or older
* Clinically evident or otherwise confirmed severe pneumonia
* SARS-CoV-2 infection confirmation (tested positive in last 14 days before randomization with locally available test system)

Exclusion Criteria:

* Known history of progressed COPD as evidenced by use of daily maintenance treatment with long-acting bronchodilators or inhaled/oral corticosteroids for > 2 months
* Patient moribund or expected to die in next 24h according to the judgment of the investigator
* Known severe congestive heart failure (New York Heart Association [NYHA] Class III- IV)
* Received organ or bone marrow transplantation in past 3 months
* Known cardio-pulmonary mechanical resuscitation in past 14 days

Phase III:

Inclusion Criteria:

* At least 18 years of age or older
* Patient on invasive mechanical ventilation (but not more than 48h post intubation at time point of first IMP administration)
* Patients with a PaO2 / FiO2 ratio of < 200 and > 60 at randomization (one representative measurement within 6h before randomization)
* SARS-CoV-2 infection confirmation (tested positive in last 14 days before randomization with locally available test system)

Exclusion Criteria:

* Intubated > 48 h at time point of first IMP administration
* Expected stop of invasive ventilation or expected extubation in the next 24h without additional intervention according to judgment of the investigator
* Known history of chronic dialysis OR received renal replacement therapy in past 14 days OR anticipated to receive renal replacement therapy within 24h after randomization
* Known history of progressed COPD as evidenced by use of daily maintenance treatment with long-acting bronchodilators or inhaled/oral corticosteroids for > 2 months
* Treatment of COVID-19 with investigational antibody treatment(s) which are not approved or not included in locally adopted treatment guidelines (e.g., WHO guidance, National Institutes of Health [NIH] COVID-19 treatment guidelines) for this indication in the past 7 days (Note: Antibody treatment[s] given within past 7 days for pre-existing diseases, other than COVID-19, are allowed.)
* At time point of randomization, treatment of COVID-19 with investigational treatments which are not approved or not included in locally adopted treatment guidelines for this indication (e.g., WHO guidance, NIH COVID-19 treatment guidelines), including SARS-CoV-2 multiplication inhibitor(s) or immunomodulator(s). (Note: If a locally adopted treatment guideline recommends drugs such as remdesivir, dexamethasone, or anticoagulation, this would be allowed. Adopted guidelines and updates must be documented at study initiation and throughout the conduct of the study.)
* Received cytokine adsorption therapy in past 3 days
* Known severe congestive heart failure (corresponding to e.g. NYHA Class III-IV, left ventricular ejection fraction <40%)
* Known history of chronic liver disease (Child-Pugh B or C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Vlaar, MD, PhD, Principal Investigator — University Amsterdam
Locations (48):
- Belgium (5):
  - InflaRx Site #1107, Aalst
  - InflaRx Site #1102, Brussels
  - InflaRx Site #1104, Leuven
  - InflaRx Site #1106, Lodelinsart
  - InflaRx Site #1101, Yvoir
- Brazil (7):
  - InflaRx Site #0301, Belo Horizonte
  - InflaRx Site #0302, Campinas
  - InflaRx Site #0305, Criciúma
  - InflaRx Site #0308, Curitiba
  - InflaRx Site #0304, Porto Alegre
  - InflaRx Site #0303, São José
  - InflaRx Site #0306, São Paulo
- France (10):
  - InflaRx Site #1011, Grenoble
  - InflaRx Site #1005, Nantes
  - InflaRx Site #1009, Nantes
  - InflaRx Site #1003, Nice
  - InflaRx Site #1001, Paris
  - InflaRx Site #1004, Paris
  - InflaRx Site #1006, Paris
  - InflaRx Site #1008, Paris
  - InflaRx Site #1012, Saint-Etienne
  - InflaRx Site #1002, Suresnes
- Germany (8):
  - InflaRx Site #0201, Aachen
  - InflaRx Site #0207, Augsburg
  - InflaRx Site #0202, Berlin
  - InflaRx Site #0208, Dresden
  - InflaRx Site #0204, Essen
  - InflaRx Site #0203, Greifswald
  - InflaRx Site #0205, Hanover
  - InflaRx Site #0206, Jena
- Mexico (6):
  - InflaRx Site #0502, Chihuahua City
  - InflaRx Site #0503, Culiacán
  - InflaRx Site #0506, Mérida
  - InflaRx Site #0504, Monterrey
  - InflaRx Site #0501, Nuevo León
  - InflaRx Site #0505, Veracruz
- Netherlands (5):
  - InflaRx Site #0101, Amsterdam
  - InflaRx Site #0103, Amsterdam
  - InflaRx Site #0106, Eindhoven
  - InflaRx Site #0104, Enschede
  - InflaRx Site #0102, Maastricht
- Peru (3):
  - InflaRx Site #0601, Callao
  - InflaRx Site #0603, Lima
  - InflaRx Site #0604, Lima
- Russia (3):
  - InflaRx Site #0701, Barnaul
  - InflaRx Site #0704, Moscow
  - InflaRx Site #0702, Ryazan
- InflaRx Site # 0804, Somerset West, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Amstel RBE, Slim MA, Lim EHT, Ruckinger S, Seymour CW, Burnett BP, Bos LDJ, van Vught LA, Riedemann NC, van de Beek D, Vlaar APJ; PANAMO Study Group. Heterogeneity of treatment effect of vilobelimab in COVID-19: a secondary analysis of a randomised controlled trial. Crit Care. 2024 Jun 28;28(1):210. doi: 10.1186/s13054-024-05004-z. PMID 38943192
- [Derived] Lim EHT, Vlaar APJ, de Bruin S, Ruckinger S, Thielert C, Habel M, Guo R, Burnett BP, Dickinson J, Brouwer MC, Riedemann NC, van de Beek D; PANAMO study group. Pharmacokinetic analysis of vilobelimab, anaphylatoxin C5a and antidrug antibodies in PANAMO: a phase 3 study in critically ill, invasively mechanically ventilated COVID-19 patients. Intensive Care Med Exp. 2023 Jun 19;11(1):37. doi: 10.1186/s40635-023-00520-8. PMID 37332066
- [Derived] Vlaar APJ, Witzenrath M, van Paassen P, Heunks LMA, Mourvillier B, de Bruin S, Lim EHT, Brouwer MC, Tuinman PR, Saraiva JFK, Marx G, Lobo SM, Boldo R, Simon-Campos JA, Cornet AD, Grebenyuk A, Engelbrecht JM, Mukansi M, Jorens PG, Zerbib R, Ruckinger S, Pilz K, Guo R, van de Beek D, Riedemann NC; PANAMO study group. Anti-C5a antibody (vilobelimab) therapy for critically ill, invasively mechanically ventilated patients with COVID-19 (PANAMO): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2022 Dec;10(12):1137-1146. doi: 10.1016/S2213-2600(22)00297-1. Epub 2022 Sep 7. PMID 36087611
- [Derived] Vlaar APJ, Lim EHT, de Bruin S, Ruckinger S, Pilz K, Brouwer MC, Guo RF, Heunks LMA, Busch MH, van Paassen P, Riedemann NC, van de Beek D. The anti-C5a antibody vilobelimab efficiently inhibits C5a in patients with severe COVID-19. Clin Transl Sci. 2022 Apr;15(4):854-858. doi: 10.1111/cts.13213. Epub 2022 Jan 14. PMID 35029045
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Vlaar APJ, de Bruin S, Busch M, Timmermans SAMEG, van Zeggeren IE, Koning R, Ter Horst L, Bulle EB, van Baarle FEHP, van de Poll MCG, Kemper EM, van der Horst ICC, Schultz MJ, Horn J, Paulus F, Bos LD, Wiersinga WJ, Witzenrath M, Rueckinger S, Pilz K, Brouwer MC, Guo RF, Heunks L, van Paassen P, Riedemann NC, van de Beek D. Anti-C5a antibody IFX-1 (vilobelimab) treatment versus best supportive care for patients with severe COVID-19 (PANAMO): an exploratory, open-label, phase 2 randomised controlled trial. Lancet Rheumatol. 2020 Dec;2(12):e764-e773. doi: 10.1016/S2665-9913(20)30341-6. Epub 2020 Sep 28. PMID 33015643

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Started | 15 | 15 | 178 | 191
Contributed to Full Analysis Set (FAS) | 15 | 15 | 177 (One patient was randomized in error and was excluded from Full Analysis Set.) | 191
Contributed to Safety Analysis Set (SAF) | 15 | 15 | 175 | 189
Completed | 13 | 11 | 103 | 93
Not Completed | 2 | 4 | 75 | 98

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (excluding one subject who was randomized in error to group Phase III: IFX-1 + SOC)
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC | Total
Number analyzed (Participants) | 15 | 15 | 177 | 191 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (8.6) | 62.8 (8.1) | 56.7 (13.2) | 55.9 (14.5) | 56.6 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 52 | 64 | 124
  Male | 11 | 11 | 125 | 127 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 8 | 11 | 115 | 119 | 253
  Race: Asian | 5 | 2 | 4 | 5 | 16
  Race: Black or African American | 2 | 2 | 5 | 8 | 17
  Race: American Indian or Alaskan Native | 0 | 0 | 22 | 24 | 46
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Multiple | 0 | 0 | 1 | 0 | 1
  Race: Other | 0 | 0 | 16 | 19 | 35
  Race: Not reported | 0 | 0 | 14 | 16 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 60 | 68 | 128
  Ethnicity: Not Hispanic or Latino | 15 | 15 | 70 | 73 | 173
  Ethnicity: Not Reported | 0 | 0 | 28 | 35 | 63
  Ethnicity: Unknown | 0 | 0 | 11 | 11 | 22
  Ethnicity: Missing | 0 | 0 | 8 | 4 | 12
Intubation status [Count of Participants; unit: Participants]
  No | 7 | 5 | 0 | 0 | 12
  Yes | 8 | 10 | 177 | 191 | 386
Oxygenation index [Mean (Standard Deviation); unit: index] — Oxygenation Index: Partial pressure of oxygen in the arterial blood (PaO2) / fractional inspired oxygen (FiO2)); Higher values indicate better health.
  index | 137.9 (51.1) | 144.2 (41.5) | 131.9 (39.2) | 130.6 (44.8) | 131.9 (42.5)

OUTCOME MEASURES:

1. Primary Outcome: Phase II: Relative Change From Baseline in Oxygenation Index in Supine Position at Day 5 (FAS)
Description: Relative change (%) from baseline in Oxygenation Index (OI; partial pressure of oxygen in the arterial blood (PaO2) / fractional inspired oxygen (FiO2)) in supine position for ≥2 hours at day 5 (FAS)
Time Frame: Baseline and Day 5
Population: Full Analysis Set (FAS) including all randomized patients according to intention-to-treat principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC
Number analyzed (Participants) | 15 | 15
percentage of change | 15.5 [-11.4 to 42.4] | 31.9 [6.0 to 57.9]
Statistical Analysis 1: Comparison: Phase II: IFX-1 + BSC vs Phase II: BSC; Test type: Superiority; p = 0.3677, Linear repeated measures model; LS means difference = -16.4, 95% CI 2-sided [-53.2 to 20.3]

2. Primary Outcome: Phase III: 28-day All-cause Mortality (FAS)
Description: Number and percentage of deaths (all-cause) until Day 28 (FAS)
Time Frame: Day 28
Population: Full Analysis Set (FAS) including all randomized patients according to intention-to-treat principle except for patients who were randomized in error AND did not receive IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Number analyzed (Participants) | 177 | 191
Participants
  Dead | 54 | 77
  Alive | 115 | 105
  Missing | 8 | 9
Statistical Analysis 1: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Cox proportional hazards regression model with outcome 28-day all-cause mortality (censored time to event variable with event = Death) including stratification by site; 61 patients from sites with no events (no death) or from single patient sites with death factually make no contribution to the analysis outcome; Test type: Superiority; p = 0.0941, Regression, Cox; including stratification by site; Hazard Ratio (HR) = 0.728, 95% CI 2-sided [0.502 to 1.056]
Statistical Analysis 2: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Cox proportional hazards regression model with outcome 28-day all-cause mortality (censored time to event variable with event = Death) without stratification by site; Post-hoc analysis; Test type: Superiority; p = 0.0266, Regression, Cox; Without stratification by site; Hazard Ratio (HR) = 0.674, 95% CI 2-sided [0.476 to 0.955]
Statistical Analysis 3: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Cox proportional hazards regression model with outcome 28-day all-cause mortality (censored time to event variable with event = Death) including random effect for site (frailty model); Post-hoc analysis; Test type: Superiority; p = 0.0181, Regression, Cox; Including random effect for site (frailty model); Hazard Ratio (HR) = 0.648, 95% CI 2-sided [0.453 to 0.929]
Statistical Analysis 4: Comparison: Phase III: IFX-1 + SOC; Cox proportional hazards regression model with outcome 28-day all-cause mortality (censored time to event variable with event = Death) including stratification by country; Post-hoc analysis; Test type: Superiority; p = 0.0067, Regression, Cox; Including stratification by country; Hazard Ratio (HR) = 0.613, 95% CI 2-sided [0.430 to 0.873]
Statistical Analysis 5: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Sensitivity analysis; 369 patients were included in this analysis including the patient that was randomized in error and not treated. Missing values were imputed by multiple imputation; Test type: Superiority; p = 0.0293, Regression, Logistic; Multiple imputation of missing values; Risk Difference (RD) = -11.0, 95% CI 2-sided [-20.8 to -1.2] — Risk difference and lower/upper limit of the Confidence Interval are given in percent
Statistical Analysis 6: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Post-hoc analysis; Test type: Superiority; p = 0.0407, Log Rank

3. Secondary Outcome: Phase II: All-cause 28-day Mortality (FAS)
Description: Number and percentage of deaths (all-cause) until Day 28 (FAS)
Time Frame: Day 28
Population: Full Analysis Set (FAS) including all randomized patients according to intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC
Number analyzed (Participants) | 15 | 15
Participants | 2 | 4
Statistical Analysis 1: Comparison: Phase II: IFX-1 + BSC vs Phase II: BSC; Cox proportional hazards regression model with outcome 28-day all-cause mortality (censored time to event variable with event = Death); Test type: Superiority; p = 0.6494, Regression, Cox; Covariate: Treatment (IFX-1 + BSC); Hazard Ratio (HR) = 0.651, 95% CI 2-sided [0.103 to 4.135]

4. Secondary Outcome: Phase II: Early Response at Day 7 After Enrollment
Description: Number of patients (%) achieving an early response at day 7 after enrollment (FAS)
Time Frame: Day 7
Population: The analysis of early response as planned in the protocol was not performed because the necessary data were not collected.
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Phase II: Late Response Until Day 28 After Enrollment
Description: Number of patients (%) reaching a late response until day 28 (FAS)
Time Frame: Baseline until Day 28
Population: The analysis of late response as planned in the protocol was not performed because the necessary data were not collected.
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Phase II: Relative Change From Baseline in Oxygenation Index in Supine Position (FAS)
Description: Relative change (%) from baseline in Oxygenation Index (OI) in supine position for ≥2 hours at days 3, 7, 9, 11, and 15 (FAS)
Time Frame: Baseline, Day 3, Day 7, Day 9, Day 11, Day 15
Population: Full Analysis Set (FAS) including all randomized patients according to intention-to-treat principle.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC
Number analyzed (Participants) | 15 | 15
percentage of change
  Day 3 | 7.1 [-10.3 to 24.4] | 17.6 [0.8 to 34.4]
  Day 7 | 13.1 [-23.4 to 49.6] | 36.0 [0.8 to 71.2]
  Day 9 | 20.7 [-15.5 to 56.9] | 27.8 [-7.2 to 62.8]
  Day 11 | 45.5 [2.1 to 88.9] | 43.5 [1.7 to 85.4]
  Day 15 | 78.5 [19.1 to 138.0] | 82.6 [25.2 to 140.0]

7. Secondary Outcome: Phase III: 60-day All-cause Mortality (FAS)
Description: Number and percentage of deaths (all-cause) until Day 60 (FAS)
Time Frame: Day 60
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Number analyzed (Participants) | 177 | 191
Participants
  Dead | 62 | 87
  Alive | 102 | 93
  Missing | 13 | 11
Statistical Analysis 1: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Cox proportional hazards regression model with outcome 60-day all-cause mortality (censored time to event variable with event = Death); Covariate: Treatment (IFX-1 + SOC); Test type: Superiority; p = 0.0815, Regression, Cox; Hazard Ratio (HR) = 0.735, 95% CI 2-sided [0.519 to 1.039]

8. Secondary Outcome: Phase III: Percentage of Patients With an Improvement in the 8-point Ordinal Scale (FAS)
Description: Percentage of patients with an improvement in the 8-point ordinal scale (Day 15, Day 28), the scale ranges from 0 = 'No clinical or virological evidence of infection' to 8 = 'Death' with higher scores meaning greater limitation and ventilation/organ support
Time Frame: Day 15, Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Number analyzed (Participants) | 177 | 191
Participants
  Improved | 82 | 77
  Not improved | 86 | 104
  Not evaluable | 9 | 10
Statistical Analysis 1: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; At Day 15; Test type: Superiority; p = 0.1553, Regression, Logistic; Risk Difference (RD) = 7.352, 95% CI 2-sided [-2.762 to 17.465] — Risk difference (IFX-1 - Placebo) of percentage of patients with an improvement in the 8-point ordinal scale; Risk difference and lower/upper limit of the CI are given in percent
Statistical Analysis 2: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; At Day 28; Test type: Superiority; p = 0.1181, Regression, Logistic; Risk Difference (RD) = 8.078, 95% CI 2-sided [-1.968 to 18.125] — [estimate comment as in outcome 8, analysis 1]

9. Secondary Outcome: Phase III: Percentage of Patients Developing Acute Kidney Failure Until Day 28 (FAS)
Description: Percentage of patients developing acute kidney failure (estimated glomerular filtration rate [eGFR] < 15 mL/min/1.73m², assessed by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] equation requiring race information) until Day 28 (FAS)
Time Frame: Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Number analyzed (Participants) | 177 | 191
Participants
  Acute kidney failure | 8 | 12
  No acute kidney failure | 158 | 168
  Not evaluable | 11 | 11
Statistical Analysis 1: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Test type: Superiority; p = 0.4105, Regression, Logistic; Risk Difference (RD) = -2.081, 95% CI 2-sided [-6.949 to 2.787] — Risk difference (IFX-1 - Placebo) of percentage of patients developing acute kidney failure; Risk difference and lower/upper limit of the CI are given in percent

10. Secondary Outcome: Phase III: Percentage of Patients Free of Any Renal Replacement Therapy Within 28 Days Upon Randomization (FAS)
Description: Percentage of patients free of any renal replacement therapy (RRT) within 28 days upon randomization (FAS), number of patients free of any RRT = number of patients - number of patients with RRT initiated after randomization until Day 28
Time Frame: Day 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC
Number analyzed (Participants) | 177 | 191
Participants | 160 | 161
Statistical Analysis 1: Comparison: Phase III: IFX-1 + SOC vs Phase III: Placebo + SOC; Test type: Superiority; p = 0.0422, Regression, Cox — p-value refers to hazard ratio from cause-specific Cox proportional hazards model for first renal replacement therapy; Covariate: Treatment (IFX-1 + SOC); Hazard Ratio (HR) = 0.539, 95% CI 2-sided [0.297 to 0.978]

ADVERSE EVENTS:
Time Frame: Phase II study part: 4 weeks; Phase III study part: 60 days;
Description: All adverse events are reported including non-treatment-emergent adverse events.
Groups:
- Phase III: IFX-1 + SOC: Phase III study part: IFX-1: 800mg intravenously administered, SOC: Standard of care; with at least one IMP administration;
- Phase III: Placebo + SOC: Phase III study part: Placebo: placebo infusion intravenously administered, SOC: Standard of care; with at least one IMP administration;
- Phase III: Randomized Non-treated Patients: Phase III study part: patients who were randomized but never treated.
Arm/Group | Phase II: IFX-1 + BSC | Phase II: BSC | Phase III: IFX-1 + SOC | Phase III: Placebo + SOC | Phase III: Randomized Non-treated Patients
All-Cause Mortality (participants affected / at risk) | 2/15 | 4/15 | 62/175 | 86/189 | 1/5
Serious Adverse Events (participants affected / at risk) | 9/15 | 7/15 | 103/175 | 122/189 | 2/5
Other Adverse Events (participants affected / at risk) | 14/15 | 14/15 | 147/175 | 154/189 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: IFX-1 + BSC (N=15) | Phase II: BSC (N=15) | Phase III: IFX-1 + SOC (N=175) | Phase III: Placebo + SOC (N=189) | Phase III: Randomized Non-treated Patients (N=5)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 21 (29) | 16 (18) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 6 (8) | 3 (3) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 24 (29) | 30 (34) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 14 (21) | 11 (14) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 9 (9) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 10 (11) | 3 (3) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 7 (7) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 6 (6) | 4 (5) | 0 (0)
Acinetobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Pneumonia acinetobacter (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Herpes simplex pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Stenotrophomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Citrobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterobacter pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nosocomial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia serratia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Tracheobronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholangitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corynebacterium sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobacter tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Morganella infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Providencia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Severe acute respiratory syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stenotrophomonas sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 12 (12) | 14 (14) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 20 (23) | 24 (25) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 7 (8) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (4) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinal shift (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary necrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 16 (16) | 31 (32) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 4 (4) | 16 (16) | 21 (21) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fibrosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Medical device site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac perforation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke in evolution (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Distributive shock (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstructive shock (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic infarction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
End-tidal CO2 increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchoalveolar lavage abnormal (Investigations) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Aspergillus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Herpes simplex test positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glutamate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sputum culture positive (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Acid-base balance disorder mixed (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive emergency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase II: IFX-1 + BSC (N=15) | Phase II: BSC (N=15) | Phase III: IFX-1 + SOC (N=175) | Phase III: Placebo + SOC (N=189) | Phase III: Randomized Non-treated Patients (N=5)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 22 (27) | 12 (16) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 8 (9) | 7 (7) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 5 (7) | 11 (13) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 7 (8) | 11 (12) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 5 (5) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 3 (3) | 11 (11) | 8 (8) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 17 (18) | 13 (13) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 7 (8) | 5 (9) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 11 (12) | 13 (15) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6) | 2 (2) | 8 (8) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 7 (9) | 8 (12) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 6 (7) | 11 (20) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 4 (4) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Refeeding syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 3 (4) | 4 (4) | 14 (15) | 13 (13) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (9) | 9 (9) | 0 (0)
Intensive care unit delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 9 (9) | 7 (7) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 10 (19) | 9 (21) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (1) | 15 (18) | 17 (31) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site vesicles (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site haemorrhage (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 3 (3) | 9 (9) | 8 (8) | 0 (0)
Blood bicarbonate increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fluid balance positive (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Blood fibrinogen increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Computerised tomogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Culture negative (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Culture urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterococcus test positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Eosinophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sputum culture positive (Investigations) | 1 (1) | 0 (0) | 4 (4) | 4 (5) | 0 (0)
Staphylococcus test positive (Investigations) | 1 (1) | 0 (0) | 5 (5) | 8 (11) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 6 (6) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 13 (13) | 20 (20) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defect conduction intraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 5 (9) | 4 (11) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 4 (4) | 7 (7) | 4 (4) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 6 (6) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (5) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (9) | 5 (6) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 10 (10) | 6 (6) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 3 (3) | 0 (0)
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 10 (10) | 5 (6) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 14 (18) | 17 (18) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 21 (22) | 15 (15) | 0 (0)
Oliguria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4 (5) | 6 (6) | 4 (4) | 5 (7) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3) | 6 (6) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral nerve lesion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pupils unequal (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device leakage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/20/NCT04333420/Prot_SAP_000.pdf